CLINICAL TRIAL: NCT01769066
Title: Random Open Exploratory Clinical Research of Sequential Gefitinib With Pemetrexed/Platinum Compare With Pemetrexed/Platinum Treatment for Advanced Non-small Cell Lung Cancer Exploratory Clinical Research
Brief Title: Clinical Value of Sequential Gefitinib With Pemetrexed/Platinum for Advanced NSCLC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, Deputy director of department of medical oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gefitinib-2009-cjh
Record Dates: First submitted 2013-01-10; First posted 2013-01-16 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed; Platinum

ARMS (2):
- Sequential Gefitinib With Pemetrexed/Platinum (Experimental): Pemetrexed IV 500 mg/m2 ，DAY2 DDP IV 75mg/m2 ，DAY1 OR CAP IV AUC 5,DAY1 Gefitinib PO. 250mg DAY3-16
  Interventions: Drug: Sequential Gefitinib With Pemetrexed/Platinum
- Pemetrexed/Platinum (Active Comparator): Pemetrexed IV 500 mg/m2 ，DAY2 DDP IV 75mg/m2 ，DAY1 OR CAP IV AUC 5,DAY1
  Interventions: Drug: Pemetrexed/Platinum

INTERVENTIONS:
Drug: Sequential Gefitinib With Pemetrexed/Platinum
  Arms: Sequential Gefitinib With Pemetrexed/Platinum
Drug: Pemetrexed/Platinum
  Arms: Pemetrexed/Platinum

SUMMARY:
The aim of this study is to explore the Clinical Value of Sequential Gefitinib With Pemetrexed/Platinum compare with Pemetrexed/Platinum for Advanced NSCLC.

DETAILED DESCRIPTION:
Patients will be randomized to 2 groups

ELIGIBILITY:
Inclusion Criteria:

1. 18~70 years
2. Patients who were diagnosed by the histologic, cytologic diagnosis of IIIb-IV non-small cell lung cancer
3. Presence of at least one index lesion measurable by CT scan or MRI
4. Ecog0-1
5. Expected life time longer than 12 weeks
6. Normal laboratory values:

   * leucocyte ≥ 4×109/L
   * neutrophil ≥ 1.5×109/L
   * platelet ≥ 100×109/L
   * Hemoglobin ≥ 10g/L
   * ALT and
   * AST ≤ 2.5×ULN (≤ 5×ULN if liver metastasis)
7. Signed written informed consent

Exclusion Criteria:

* Patients have used drugs according to protocol
* Patients were allergic to pemetrexed or cisplatin
* Patients received radiotherapy or other biological treatment 4 weeks before the trial
* Uncontrolled hydrothorax or hydropericardium
* neuropathy toxicity ≥ CTC 3
* Severe symptomatic heart disease
* Active upper gastrointestinal ulcer or digestive disfunction
* Severe infection or metabolic disfunction
* Patients with other malignant tumor
* Uncontrolled brain metastases
* Patients have accepted other clinical trials
* Female patients during their pregnant and lactation period, or patients without contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-12; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
12 weeks of non-progression rate | from the first cycle of treatment (day one) to two month after the last cycle

SECONDARY OUTCOMES:
PFS | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Overall Officials: Chang jian hua, MD,PhD, Principal Investigator — Cancer hospital Fudan University
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China